CLINICAL TRIAL: NCT03148587
Title: Medication Abortion Self-Confirmation (MASC): Comparison of Two Home Pregnancy Tests as an Alternative to Office Follow-up
Brief Title: Medical Abortion Self-Confirmation (MASC)
Acronym: MASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 39816
Record Dates: First submitted 2017-04-27; First posted 2017-05-11 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Medical Abortion
Keywords: abortion; medical abortion; mifepristone; pregnancy test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-level pregnancy test (MLPT) (Experimental): Patients randomized to multi-level pregnancy test (MLPT) arm will receive MLPTs to perform at home one and two weeks after taking mifepristone. They will be asked to interpret the results of the MLPT as it relates to their pregnancy termination status.
  Interventions: Behavioral: Self-assessment: MLPT
- Low sensitivity pregnancy test (LSPT) (Experimental): Patients randomized to low sensitivity pregnancy test (LSPT) arm will receive LSPTs to perform at home at one and two weeks after taking mifepristone. They will be asked to interpret the results of the LSPT as it relates to their pregnancy termination status.
  Interventions: Behavioral: Self-assessment: LSPT

INTERVENTIONS:
Behavioral: Self-assessment: MLPT — Patients enrolled in the study will self-assess the outcomes of their medical abortion using the multi-level pregnancy test.
  Arms: Multi-level pregnancy test (MLPT)
Behavioral: Self-assessment: LSPT — Patients enrolled in the study will self-assess the outcomes of their medical abortion using the low sensitivity pregnancy test.
  Arms: Low sensitivity pregnancy test (LSPT)

SUMMARY:
This study aims to investigate the ability of participants to perform and accurately interpret the multi-level pregnancy test and the low sensitivity pregnancy test following medication abortion, without routine provider contact.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of less than or equal to 63 days
* English speaking
* Determined by the site investigator or designee to be fully eligible for medical abortion with mifepristone followed by misoprostol according to the site's standard criteria
* In the judgement of the site investigator, she is capable of giving informed consent and she has signed the study informed consent or assent form

Exclusion Criteria:

* Allergy to mifepristone and/or misoprostol
* Non-english speaking
* Inability to access internet

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Correct interpretation of pregnancy test | 4 weeks after taking medication abortion medication, mifepristone

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Health Care, Stanford, California, United States